CLINICAL TRIAL: NCT03596749
Title: The Effect of Sevelamer Carbonate on Serum Trimethylamine-n-Oxide (TMAO) Level in Patients With Chronic Kidney Disease (CKD) Stage 3b-4: a Protocol of a Randomized, Parallel, Controlled Trial
Brief Title: The Effect of Sevelamer Carbonate on Serum Trimethylamine-n-Oxide (TMAO) Level in Patients With Chronic Kidney Disease (CKD) Stage 3b-4
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fan Fan Hou (Other)
Responsible Party: Sponsor-Investigator, Fan Fan Hou, Chief of Division of Nephrology, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMON
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: CKD Stage 3b; CKD Stage 4
MeSH Terms: interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevelamer Carbonate (Experimental): Sevelamer carbonate will be given with fixed dose of 1600mg (p.o. b.i.d) with meals
  Interventions: Drug: Sevelamer Carbonate
- Control (No Intervention): blank-control

INTERVENTIONS:
Drug: Sevelamer Carbonate — Sevelamer carbonate 1600mg (p.o. b.i.d) with meals
  Arms: Sevelamer Carbonate

SUMMARY:
The aim of this study is to investigate effects of sevelamer carbonate on reducing TMAO in stage 3b-4 CKD (pre-dialysis) patients. The study will also investigate the safety and tolerability of sevelamer carbonate in study population and the effects of sevelamer carbonate on serum p-cresyl sulfate, indoxyl sulfate, LDL-C and uric acid.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or women, aged from 18 to 75 years old;
* 2. Provide informed consent prior to enrolling in the study;
* 3. Estimated glomerular filtration rate (eGFR) between 15-45 ml/min/1.73 m2 (calculated by CKD-EPI equation)

Exclusion Criteria:

* 1. Documented poorly controlled diabetes mellitus, poorly controlled hypertension, malignant tumour, or any clinically significant unstable medical condition;
* 2. Active dysphagia or swallowing disorder; or a predisposition to or current bowel obstruction, ileus, or severe gastrointestinal motility disorders including severe constipation;
* 3. Known hypersensitivity to sevelamer or any constituents of the study drug;
* 4. Unable to comply with the requirements of the study;
* 5. Hypophosphatemia (serum phosphorus level <0.87mmol/L);
* 6. Women who have a positive pregnancy test at enrollment or women who are breast-feeding;
* 7. Have been enrolled in other interventional study;
* 8. Received sevelamer or other intestinal adsorbents, or broad-spectrum antibiotic within one month prior to the screening period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the serum concentration of TMAO between treatment group and control group | 22 weeks
  The serum concentration of TMAO will be evaluated by high performance liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Difference in the serum concentration of p-cresyl sulfate between treatment group and control group | 22 weeks
  The serum concentration of p-cresyl sulfate will be evaluated by high performance liquid chromatography (HPLC)
Difference in the serum concentration of indoxyl sulfate between treatment group and control group | 22 weeks
  The serum concentration of indoxyl sulfate will be evaluated by high performance liquid chromatography (HPLC)
Difference in the serum concentration of LDL-C between treatment group and control group | 22 weeks
  Chemistry evaluations
Difference in the serum concentration of uric acid between treatment group and control group | 22 weeks
  Chemistry evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Fan Fan Hou, M.D.,PhD, Principal Investigator — Division of nephrology, Nanfang Hospital Southern Medical University
Locations (1):
- Renal Division, Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Goto S, Yoshiya K, Kita T, Fujii H, Fukagawa M. Uremic toxins and oral adsorbents. Ther Apher Dial. 2011 Apr;15(2):132-4. doi: 10.1111/j.1744-9987.2010.00891.x. Epub 2011 Mar 8. PMID 21426503
- [Background] Tang WH, Wang Z, Kennedy DJ, Wu Y, Buffa JA, Agatisa-Boyle B, Li XS, Levison BS, Hazen SL. Gut microbiota-dependent trimethylamine N-oxide (TMAO) pathway contributes to both development of renal insufficiency and mortality risk in chronic kidney disease. Circ Res. 2015 Jan 30;116(3):448-55. doi: 10.1161/CIRCRESAHA.116.305360. Epub 2014 Nov 5. PMID 25599331
- [Background] Yubero-Serrano EM, Woodward M, Poretsky L, Vlassara H, Striker GE; AGE-less Study Group. Effects of sevelamer carbonate on advanced glycation end products and antioxidant/pro-oxidant status in patients with diabetic kidney disease. Clin J Am Soc Nephrol. 2015 May 7;10(5):759-66. doi: 10.2215/CJN.07750814. Epub 2015 Feb 20. PMID 25710801
- [Background] Vlassara H, Uribarri J, Cai W, Goodman S, Pyzik R, Post J, Grosjean F, Woodward M, Striker GE. Effects of sevelamer on HbA1c, inflammation, and advanced glycation end products in diabetic kidney disease. Clin J Am Soc Nephrol. 2012 Jun;7(6):934-42. doi: 10.2215/CJN.12891211. Epub 2012 Mar 29. PMID 22461535
- [Background] Rastogi A. Sevelamer revisited: pleiotropic effects on endothelial and cardiovascular risk factors in chronic kidney disease and end-stage renal disease. Ther Adv Cardiovasc Dis. 2013 Dec;7(6):322-42. doi: 10.1177/1753944713513061. PMID 24327730
- [Background] Koopen AM, Groen AK, Nieuwdorp M. Human microbiome as therapeutic intervention target to reduce cardiovascular disease risk. Curr Opin Lipidol. 2016 Dec;27(6):615-622. doi: 10.1097/MOL.0000000000000357. PMID 27676197
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117